CLINICAL TRIAL: NCT00465543
Title: A Double-blind,Placebo-controlled, Randomized, Crossover Trial of Mint Tea High in Rosmarinic Acid in Adults With Nasal Polyposis
Brief Title: Mint Tea for the Treatment of Nasal Polyps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Paul Keith, Associate Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07-010
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Nasal Polyps
Keywords: Nasal polyposis; Mint tea; Double-blind; Placebo-controlled; Crossover
MeSH Terms: conditions — Nasal Polyps | interventions — Rosmarinic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- II (Placebo Comparator): Arm 2 receives 4 weeks of placebo mint tea (consumed twice a day) followed by 4 weeks of washout and then a further 4 weeks of treatment with study mint tea (consumed twice a day).
  Interventions: Other: Mint tea low in rosmarinic acid
- I (Placebo Comparator): Arm 1 receives 4 weeks of treatment with mint tea high in rosmarinic acid, consumed twice a day. Treatment is followed by a 4 week wash-out phase. Subjects then enter a 4 week phase of placebo mint tea (low in rosmarinic acid), to be consumed twice a day.
  Interventions: Other: Mint tea high in rosmarinic acid

INTERVENTIONS:
Other: Mint tea high in rosmarinic acid — Mint tea high in rosmarininc acid contains 150mg of rosmarinic acid. To be consumed twice a day for 4 weeks. Brewed in 150ml of boiling water and allowed to steep for 10 minutes.
  Arms: I
Other: Mint tea low in rosmarinic acid — Mint tea low in rosmarininc acid contains 10mg of rosmarinic acid. To be consumed twice a day for 4 weeks. Brewed in 150ml of boiling water and allowed to steep for 10 minutes.
  Arms: II

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a new treatment for nasal polyps as compared to placebo (an inactive substance). The treatment involved is mint tea high in rosmarinic acid. Rosmarinic acid is a polyphenol, or a chemical substance found in certain plants such as oregano, rosemary, and the mints. It is the active ingredient in spearmint. The placebo used in this study will be mint tea low in rosmarininc acid. In this trial the amount of rosmarinic acid in the high rosmarinic acid tea, or study tea, will be 150mg. The placebo, or low rosmarinic acid tea, will contain 10mg of rosmarinic acid.

DETAILED DESCRIPTION:
Nasal polyps are clear, glistening, grape-like structures that occur in two percent of adults and contain a large number of activated eosinophils - about 20% of the constituents of nasal polyp tissue.

The standard treatment for nasal polyp patients is intranasal steroids which, in troublesome cases, may follow a short course of oral steroids. Surgery is reserved for extremely large polyps and those who fail medical treatment. However, many patients tire of using nasal sprays or are troubled by side effects such as nasal irritation or bleeding. So, while all treatments offer some benefit, there is no gold standard.

Rosmarinic acid is categorized as a polyphenolia phytochemical, or a 'plant phenol' and is found in a variety of plants including the herbs oregano and rosemary, as well as the mints. Peppermint is one of the most widely used single ingredient in herbal teas. It has been found in vitro to have significant antimicrobial and antiviral properties, strong antioxidant and antitumor actions, and some antiallergenic ability. Human based research is limited.

A mint tea high in rosmarinic acid has recently been produced. Anecdotal evidence suggests that it may be beneficial for allergic rhinitis if taken prior to allergen exposure (personal communication). Other anecdotal evidence found a blunting of the sputum eosinophils following allergen challenge in allergic asthmatics (personal communication). This trial aims to study the effects of this mint tea high in rosmarinic acid in adults with bilateral nasal polyps, a condition characterized by chronic eosinophilic inflammation. The control treatment will be a mint tea low in rosmarinic acid.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are male or female aged 18 years or older.
2. Subjects who have signed an informed consent agreement.
3. Subjects with a history of nasal polyp symptoms during the previous 12 months.

Exclusion Criteria:

1. Subjects with severe nasal polyps requiring immediate surgery.
2. Subjects presenting with unilateral polyps.
3. Subjects who have undergone surgery to treat their nasal polyps (nasal polypectomy) within one year prior to visit one.
4. Subjects who have a known fungal infection of the nose and/or paranasal sinuses, nasal candidiasis, acute or chronic infectious sinusitis of viral or bacterial nature.
5. Subjects who have had an upper respiratory tract infection within two weeks prior to Visit one or any time between Visit 1 and Visit 2.
6. Subjects having cystic fibrosis, Young's syndrome, primary ciliary dyskinesia, known HIV infection or alcohol abuse.
7. Subjects with clinically significant, uncontrolled evidence of cardiovascular, neurological, hepatic, renal, respiratory, or any other medical condition that may interfere with the study.
8. Subjects with a recent history (within six months) of a clinically significant psychiatric disorder other than mild depression.
9. Subjects who have any clinically relevant deviation from normal in the general physical examination.
10. Subjects who have received any depot, systemic or oral corticosteroid in the previous three months prior to the start of the study.
11. Subjects who are unable to cease treatment with intranasal steroids four weeks prior to Visit one.
12. Subjects with a known hypersensitivity to mint.
13. Females who are pregnant or lactating or are likely to become pregnant during the study or are less than 8 weeks postpartum. Women of childbearing age may be included if in the opinion of the investigator, they are taking adequate contraceptive measures.
14. Subjects who are unable to follow the instructions within this protocol or known inability to attend all clinic visits within the intervals stated.
15. Subjects who have participated in a clinical trial involving an investigational or marketed drug within four weeks of visit one.
16. Subjects who are allergy skin test positive to a seasonal allergen which will be present when performing the trial, that has caused, within the past 2 years, a clinically significant deterioration in nasal symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Nasal polyposis quality of life questionnaire | Visits 2, 3,4,5
Nasal patency as assessed by use of the Clement-Clarke peak nasal inspiratory flow meter (PNIF) | Daily

SECONDARY OUTCOMES:
Nasal lavage eosinophils. | Visits 1,2,3,4,5
Peripheral blood eosinophils | Visits 2,3,4,5
Diary symptom scores. | Daily
Nasal polyp size on visual inspection. | Visits 1,2,3,4,5
Subjects Global Assessment of symptoms | Visits 3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Paul K. Keith, Principal Investigator — Hamilton Health Sciences Corporation, McMaster Site

REFERENCES:
- [Background] Finotto S, Dolovich J, Denburg JA, Jordana M, Marshall JS. Functional heterogeneity of mast cells isolated from different microenvironments within nasal polyp tissue. Clin Exp Immunol. 1994 Feb;95(2):343-50. doi: 10.1111/j.1365-2249.1994.tb06535.x. PMID 7508349
- [Background] McKay DL, Blumberg JB. A review of the bioactivity and potential health benefits of peppermint tea (Mentha piperita L.). Phytother Res. 2006 Aug;20(8):619-33. doi: 10.1002/ptr.1936. PMID 16767798
- [Background] Takano H, Osakabe N, Sanbongi C, Yanagisawa R, Inoue K, Yasuda A, Natsume M, Baba S, Ichiishi E, Yoshikawa T. Extract of Perilla frutescens enriched for rosmarinic acid, a polyphenolic phytochemical, inhibits seasonal allergic rhinoconjunctivitis in humans. Exp Biol Med (Maywood). 2004 Mar;229(3):247-54. doi: 10.1177/153537020422900305. PMID 14988517
- [Background] Ruhno J, Andersson B, Denburg J, Anderson M, Hitch D, Lapp P, Vanzieleghem M, Dolovich J. A double-blind comparison of intranasal budesonide with placebo for nasal polyposis. J Allergy Clin Immunol. 1990 Dec;86(6 Pt 1):946-53. doi: 10.1016/s0091-6749(05)80158-7. PMID 2262649
- [Background] Keith PK, Conway M, Dolovich J. Development and validation of a nasal polyposis quality of life questionnaire. J Allergy Clin Immunol 1996;97:192(Abstract)
- [Background] Keith PK, Ferrie P, Conway M, Waserman S, Schmuck ML, Denburg JA. A double-blind, placebo-controlled, randomized, crossover trial of montelukast in adults with nasal polyposis. Allergy Clin Immunol Int: J World Allergy Org, 2003; Supp 1:185.(Abstract)
- [Background] Powell KR, Shorr R, Cherry JD, Hendley JO. Improved method for collection of nasal mucus. J Infect Dis. 1977 Jul;136(1):109-11. doi: 10.1093/infdis/136.1.109. PMID 886201